CLINICAL TRIAL: NCT06450366
Title: A Phase 3, Randomized, Double-Blind Study to Evaluate the Efficacy and Safety of MK-0616 Compared With Ezetimibe or Bempedoic Acid or Ezetimibe and Bempedoic Acid in Adults With Hypercholesterolemia
Brief Title: A Study to Evaluate the Efficacy and Safety of Enlicitide Decanoate (MK-0616, Oral PCSK9 Inhibitor) Compared With Ezetimibe or Bempedoic Acid or Ezetimibe and Bempedoic Acid in Adults With Hypercholesterolemia (MK-0616-018) CORALreef AddOn
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0616-018; MK-0616-018 (Other: MSD); 2023-504920-25 (Registry Identifier: EU CT); U1111-1290-3888 (Registry Identifier: UTN)
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-04

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — MK-0616; Ezetimibe; 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Enlicitide Decanoate (Experimental): Participants receive enlicitide decanoate 20mg, ezetimibe-matching placebo, and bempedoic acid-matching placebo once daily (QD) orally up to approximately 56 days.
  Interventions: Drug: Enlicitide Decanoate; Other: Placebo for Ezetimibe; Other: Placebo for Bempedoic Acid
- Ezetimibe (Active Comparator): Participants receive ezetimibe 10mg, enlicitide decanoate-matching placebo, and bempedoic acid-matching placebo QD orally up to approximately 56 days.
  Interventions: Drug: Ezetimibe; Other: Placebo for Enlicitide Decanoate; Other: Placebo for Bempedoic Acid
- Bempedoic Acid (Active Comparator): Participants receive bempedoic acid 180mg, ezetimibe-matching placebo, and enlicitide decanoate-matching placebo QD orally up to approximately 56 days.
  Interventions: Drug: Bempedoic Acid; Other: Placebo for Enlicitide Decanoate; Other: Placebo for Ezetimibe
- Ezetimibe + Bempedoic Acid (Active Comparator): Participants receive ezetimibe 10 mg, bempedoic acid 180mg, enlicitide decanoate-matching placebo orally QD for approximately 56 days.
  Interventions: Drug: Ezetimibe; Drug: Bempedoic Acid; Other: Placebo for Enlicitide Decanoate

INTERVENTIONS:
Drug: Enlicitide Decanoate — Administered orally.
  Other Names: MK-0616
  Arms: Enlicitide Decanoate
Drug: Ezetimibe — Administered orally.
  Arms: Ezetimibe; Ezetimibe + Bempedoic Acid
Drug: Bempedoic Acid — Administered orally.
  Arms: Bempedoic Acid; Ezetimibe + Bempedoic Acid
Other: Placebo for Enlicitide Decanoate — Administered orally.
  Arms: Bempedoic Acid; Ezetimibe; Ezetimibe + Bempedoic Acid
Other: Placebo for Ezetimibe — Administered orally.
  Arms: Bempedoic Acid; Enlicitide Decanoate
Other: Placebo for Bempedoic Acid — Administered orally.
  Arms: Enlicitide Decanoate; Ezetimibe

SUMMARY:
The main purpose of this study is to assess whether enlicitide decanoate is superior to ezetimibe or bempedoic acid or ezetimibe + bempedoic acid in reducing LDL-C in participants with hypercholesterolemia, and to evaluate its safety and tolerability. The primary study hypotheses are enlicitide decanoate is superior to ezetimibe, bempedoic acid, and ezetimibe + bempedoic acid on mean percent change from baseline in LDL-C at week 8.

ELIGIBILITY:
Inclusion Criteria:

* Has either a) history of a major atherosclerotic cardiovascular disease (ASCVD) event or b) if no history of a major ASCVD event, has intermediate to high risk for development of a first major ASCVD event
* Has fasted lipid values (evaluated by the central laboratory) at Visit 1 (Screening) as follows: a) history of a major ASCVD event with LDL-C ≥55 mg/dL (≥1.42 mmol/L) OR b) No history of a major ASCVD event with LDL-C ≥70 mg/dL (≥1.81 mmol/L)
* Is treated with a low, moderate, or high intensity statin (±non-statin lipid lowering therapy [LLT])
* Is on a stable dose of all background LLTs with no planned medication or dose changes during the study
* Is an individual of any sex/gender, from 18 years of age inclusive, at the time of providing the informed consent

Exclusion Criteria:

* Has a history of homozygous familial hypercholesterolemia (FH) based on genetic or clinical criteria, compound heterozygous familial hypercholesterolemia (HeFH), or double HeFH
* Has New York Heart Association class IV heart failure, or last known left ventricular ejection fraction ≤25% by any imaging method, or had a heart failure hospitalization within 3 months before Visit 1 (Screening)
* Participants with a history of tendon disorder or tendon rupture
* Participants with a history of gout
* Is undergoing or previously underwent an LDL-C apheresis program within 3 months before Visit 1 (Screening) or plans to initiate an LDL-C apheresis program
* Was previously treated/is being treated with certain other cholesterol lowering medications, including ezetimibe, bempedoic acid, or protein convertase subtilisin/kexin type 9 (PCSK9) inhibitors without adequate washout

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Mean Percent Change from Baseline in LDL-C at Day 56 | Baseline and Day 56
  Blood samples will be collected at baseline and after 56 days of treatment to assess mean percentage change in LDL-C. The percent change from baseline in LDL-C at Day-56 will be reported.

SECONDARY OUTCOMES:
Mean Percent Change from Baseline in Apolipoprotein B (ApoB) at Day 56 | Baseline and Day 56
  Blood samples will be collected at baseline and on day 56 of treatment to assess mean percent change in ApoB. The percent change from baseline in ApoB at Day 56 will be reported.
Mean Percent Change from Baseline in Non-High-density Lipoprotein Cholesterol (Non-HDL-C) at Day 56 | Baseline and Day 56
  Blood samples will be collected at baseline and on day 56 of treatment to assess mean percent change in non-HDL-C. The percent change from baseline in non-HDL-C at 56 days will be reported.
Percent Change from Baseline in Lipoprotein(a) Levels (Lp[a]) | Baseline and Day 56
  Blood samples will be collected at baseline and on day 56 of treatment to assess percent change in Lp(a) levels. The change from baseline at Day 56 will be reported.
Percentage of Participants Who at Day 56 Have an LDL-C <70 mg/dL and ≥50% Reduction from Baseline | Baseline and Day 56
  The percentage of participants who have an LDL-C <70 mg/dL and >50% reduction from baseline at day 56 will be reported.
Percentage of Participants Who at Day 56 Have an LDL-C <55 mg/dL and ≥50% Reduction from Baseline | Baseline and Day 56
  The percentage of participants who have an LDL-C <55 mg/dL and >50% reduction from baseline at day 56 will be reported.
Number of Participants With ≥1 Adverse Event (AE) | Up to Approximately 112 days
  An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Number of Participants Discontinuing from Study Therapy Due to AE | Up to Approximately 56 days
  An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (35):
- United States (7):
  - Clinical Trials Research ( Site 1509), Lincoln, California
  - Healthcare Research Network - Chicago ( Site 1507), Flossmoor, Illinois
  - L-MARC Research Center ( Site 1501), Louisville, Kentucky
  - Velocity Clinical Research Rockville ( Site 1503), Rockville, Maryland
  - Velocity Clinical Research, Gulfport ( Site 1505), Gulfport, Mississippi
  - Piedmont Research Partners ( Site 1506), Fort Mill, South Carolina
  - Rainier Clinical Research Center ( Site 1502), Renton, Washington
- Argentina (3):
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 1002), Mar del Plata, Buenos Aires
  - CIPREC-CIPREC Sede Arenales ( Site 1000), Buenos Aires, Buenos Aires F.D.
  - Fundacion Estudios Clinicos ( Site 1001), Rosario, Santa Fe Province
- Canada (5):
  - The Medical Arts Health Research Group ( Site 1606), Vancouver, British Columbia
  - Cambridge Cardiac Care Centre ( Site 1603), Cambridge, Ontario
  - North York Diagnostic and Cardiac Centre ( Site 1605), North York, Ontario
  - Institut de Cardiologie de Montreal ( Site 1604), Montreal, Quebec
  - Diex Recherche Trois-Rivieres ( Site 1602), Trois-Rivières, Quebec
- France (4):
  - Hôpital Arnaud de Villeneuve - CHU Montpellier ( Site 0505), Montpellier, Herault
  - Hôpital Nord Guillaume-et-René-Laennec / CHU de Nantes-CIC Endocrinology-Diabetology-Nutrition ( Sit, Nantes, Loire-Atlantique
  - Hospices Civils de Lyon - Hopital Louis Pradel ( Site 0501), Bron, Rhone
  - Hôpital Bichat - Claude-Bernard ( Site 0504), Paris
- Israel (4):
  - Yitzhak Shamir Medical Center. ( Site 0702), Beer Yaakov
  - Assuta Beersheba MC ( Site 0704), Beersheba
  - Rambam Health Care Campus ( Site 0700), Haifa
  - Meir Medical Center. ( Site 0703), Kfar Saba
- Spain (5):
  - Hospital Universitario Virgen de la Victoria-UGC Endocrinologia y nutricion ( Site 0801), Málaga, Andalusia
  - Hospital de Figueres ( Site 0804), Figueres, Gerona
  - Hospital San Rafael de Coruna ( Site 0805), A Coruña, La Coruna
  - EAP Sardenya ( Site 0800), Barcelona
  - Hospital Universitari Vall d'Hebron ( Site 0803), Barcelona
- Taiwan (4):
  - National Cheng Kung University Hospital-Internal Medicine ( Site 0403), Tainan
  - National Taiwan University Hospital ( Site 0400), Taipei
  - Taipei Veterans General Hospital-Department of Medicine ( Site 0402), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 0404), Taoyuan District
- United Kingdom (3):
  - Barts Health NHS Trust-William Harvey Clinical Research Centre ( Site 0901), London, England
  - Royal Free Hospital ( Site 0900), London, England
  - National Institute for Health Research UCLH Clinical Research Facility ( Site 0908), London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26302&tenant=MT_MSD_9011